CLINICAL TRIAL: NCT03295760
Title: Analysis of Q10 Coenzyme Efficacy for Long-term Treatment of Cyclic Vomiting Syndrome in Children
Acronym: COENZYME
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/COENZYME-FEILLET/VS
Record Dates: First submitted 2017-09-21; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Cyclic Vomiting Syndrome
MeSH Terms: conditions — Familial cyclic vomiting syndrome | interventions — Ubiquinone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cyclic vomiting syndrome: Children followed at Children's Hospital of Nancy treated with Q10 coenzyme for cyclic vomiting syndrome
  Interventions: Drug: Q10 Coenzyme

INTERVENTIONS:
Drug: Q10 Coenzyme

SUMMARY:
The main purpose of this study is the comparison of frequency of vomiting episodes (number of episodes per year) observed during the year after the begin of Q10 coenzyme treatment to frequency observed during the year before the begin of this treatment in children with cyclic vomiting syndrome.

Secondary purposes are the evaluation of life quality of parents and children, of treatment safety and its economic cost compared to other recommended treatments.

ELIGIBILITY:
Inclusion Criteria:

* Cyclic vomiting syndrome as defined by Rome IV criteria
* Treated with Q10 coenzyme treatment for cyclic vomiting syndrome
* Q10 coenzyme treatment started between January 2000 and July 2006

Exclusion Criteria:

- Refusal of processing of personal data reported in patient medical files

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children followed at Children's Hospital of Nancy treated with Q10 coenzyme for cyclic vomiting syndrome
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of vomiting episodes | from date of inclusion (start of Q10 coenzyme treatment) up to 1 year
  measured by number of episodes per year
Frequency of vomiting episodes | from 1 year before date of inclusion until date of inclusion (start of Q10 coenzyme treatment)
  measured by number of episodes per year

SECONDARY OUTCOMES:
Intensity of vomiting episodes | from 1 year before date of inclusion until date of inclusion (start of Q10 coenzyme treatment)
  reported by the child and/or parents
Intensity of vomiting episodes | from date of inclusion (start of Q10 coenzyme treatment) up to 1 year
  reported by the child and/or parents
Number of child hospitalizations | from 1 year before date of inclusion until date of inclusion (start of Q10 coenzyme treatment)
Number of child hospitalizations | from date of inclusion (start of Q10 coenzyme treatment) up to 1 year
Cost of Q10 coenzyme treatment and other recommended treatments for cyclic vomiting syndrome | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital - CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No